CLINICAL TRIAL: NCT06141772
Title: Prospective Study of Circulating Tumor DNA Kinetics Post R-CHOP Type Treatment of Diffuse Large B Cell Lymphoma
Brief Title: Kinetics of Circulating Tumor DNA in Lymphoma Treated by Immuno-chemotherapy
Acronym: LYMPHO-CLEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB23.05
Record Dates: First submitted 2023-10-17; First posted 2023-11-21 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse Large B Celle Lymphoma; Circulating tumor DNA
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kinetics of circulating tumor DNA (Experimental)
  Interventions: Other: Measure of the circulating tumor DNA

INTERVENTIONS:
Other: Measure of the circulating tumor DNA — Blood assessment to measure the kinetics au circulating tumor DNA

SUMMARY:
The purpose of this study is to determine the kinetics of circulating tumor DNA (ctDNA) in the hours following initial administration of immuno-chemotherapy to patients with diffuse large B cell lymphoma (DLBCL). Modelizing the short-term kinetics of ctDNA would help to determine the optimal time-point for ctDNA follow-up. The investigators hypothesize that the greater ctDNA release at this time-point compared to baseline might lead lead to the detection of novel variants compared to baseline.

DETAILED DESCRIPTION:
ctDNA in diffuse large B cell lymphoma (DLBCL) has become an essential dynamic biomarker. Due to its short half-life, ctDNA is a real-time reflection of tumoral evolution and is a non-invasive biomarker that can be used for patient evaluation and follow-up. The quantity of ctDNA before treatment is correlated with tumoral mass, international prognostic index (IPI) and prognosis. The principal mechanism of ctDNA release is tumor cell apoptosis and it is well established that tumor cell apoptosis is observed in the hours following immuno-chemotherapy. However, the kinetics of ctDNA concentration in the hours following immuno-chemotherapy administration is unknown.

Modelizing the kinetics of ctDNA during this early timeframe could help to better predict chemo-sensitivity and better reflect genetic heterogeneity of the tumor, through release of a larger quantity of ctDNA compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diffuse Large B Cell Lymphoma
* TEP-TDM at diagnosis
* Inform Consent form signed
* Performance status 0 or 1
* Hospitalized on clinician decision for first cycle of R-CHOP or R-miniCHOP

Exclusion Criteria:

* Histology other than Diffuse Large B Cell
* Patient under guardianship or curatorship
* Incapacity to understand the study or conform to the constraints of the study (language barrier, psychological barrier, geographic barrier…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Analysis of circulating tumor DNA kinetics | 21 days
  Blood assessment to measure circulating tumor concentration

SECONDARY OUTCOMES:
Correlation between circulating tumor DNA concentration and metabolic volume | 6 months
  comparison between circulating tumoral concentration and metabolic volume measured on TEP

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Jardin, MD,PhD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France